CLINICAL TRIAL: NCT04345731
Title: Over-the-counter (OTC) Labels for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Mark Becker, Professor Department of Psychology, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000832
Record Dates: First submitted 2020-04-01; First posted 2020-04-14 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Adverse Drug Event
Keywords: drug labels
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Several different studies within one large study to explore the use of over the counter medical labels and reducing adverse side effects. Each study is a repeated subjects design, with each participant receiving all label treatments to allow a within subjects analysis of label effectiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1 - Control (No Intervention): We note that our within subjects experimental design, in which each subject receives all treatments, is not well suited to this system of reporting. Thus we are defining "arms" as the label treatments we are evaluating. This label is the control label treatment which represents the current, legally required over-the-counter labeling standard.
- Condition 2 - Highlighted (Experimental): This condition will involve a novel method of presenting critical active ingredient, drug/drug, and drug/diagnosis information with highlighting.
  Interventions: Other: Over the counter drug labels
- Condition 3 - FOP warning label (Experimental): This condition will involve presenting critical drug/drug, and drug/diagnosis information in a novel Front-of-Pack (FOP) warning label.
  Interventions: Other: Over the counter drug labels
- Condition 4- FOP+Highlighting label (Experimental): This condition will combine both the highlighting and FOP labeling interventions from conditions 2 and 3. Note: Across the four arms we are essentially doing a 2 (highlighting/no highlighting) by 2 (front of pack warning/ no front of pack warning) within subjects design.
  Interventions: Other: Over the counter drug labels

INTERVENTIONS:
Other: Over the counter drug labels — A control condition based on the current standard OTC label and 3 experimental labels will be compared to identify OTC labels that more effectively communicate critical information for the reduction of adverse drug events to the consumer
  Other Names: OTC drug label
  Arms: Condition 2 - Highlighted; Condition 3 - FOP warning label; Condition 4- FOP+Highlighting label

SUMMARY:
Optimizing OTC labels for older adults: Empirical evaluation of labels designed to provide older users the information they need to to minimize adverse drug events

DETAILED DESCRIPTION:
The overarching goal is to design and evaluate a novel front of pack label for OTC drugs that will reduce the prevalence of Adverse Drug Reactions (ADRs) in older adults. To do so the researchers will survey pharmacists to ascertain which label information is most important to the reduction of ADRs, and then will design novel OTC labels which highlight this information. To evaluate the effectiveness of these designs, the investigators propose five experiments where older adults will make judgments about OTC appropriateness.

Study 1 - Survey of Pharmacists - Overseen by University of Wisconsin - Online Survey of pharmacists to evaluate which aspects in a drug facts labels are most critical to the reduction of adverse drug events.

Experiment 2 - Change Detection- Computer screen flashes between a label and the same label which has been modify slightly. Participant is instructed to locate the change as quickly as possible. Change should be detected more quickly for labels that engage users in bottom-up processing.

Experiment 3A- Absolute Judgement- Participant is asked a yes/no question about whether a product being displayed on a computer monitor is appropriate given a scenario. Half the scenarios involve active ingredient and half warning information. Time accuracy will indicate which labels are most effective.

Experiment 3B-Cross Product Comparison-Participant is given a scenario (that requires active ingredient or warning information) and is asked to select the appropriate OTC from a set of options(both products presented in identical labeling format within a trial). Again, speed an accuracy will be used to evaluate the most effective label designs.

Experiment 4- Judging Product Appropriateness- Participants judge whether a drug is appropriate for them based on their health and current medications. Information content varies across trials to determine how much information is required to make an informed decision. Response accuracy (relative to expert pharmacists from the University of Wisconsin's evaluation) as a function of the information presented will be used to determine information that is critical to make a correct decision and how well do the participants get that information from the standard principle display panel (PDP- the front panel) and the Drug Facts Label.

Experiment 5 - Eye tracking during appropriateness judgments - Participants evaluate whether an OTC medication is appropriate for their use, given their current health status and medication intake. Label formats will include current standards and an optimized label (derived from earlier experiments). Appropriateness judgments will be evaluated by pharmacists at University of Wisconsin, and the participant's eye movements will be monitored as they inspect the drugs. Comparisons across drug label formats will allow the primary investigators at Michigan State University to evaluate whether the optimized format more effectively garners attention and improves decision making.

Experiment 6 - Will be a replication of Experiment 5's methods but will use commercial brands rather than the mock brands in Experiment 5. This will allow the primary investigators at Michigan State University to evaluate the extent to which the effects found in Experiment 5 generalize to commercial brands about which participants may have prior familiarity and which contain branding information.

ELIGIBILITY:
Inclusion Criteria:

* participant must be 65+
* participant must be legally sighted
* participant must be able purchase and administer their own medications
* participant must be able to perform consent without assistance.

Exclusion Criteria:

* if the participant has history of seizures
* if the participant has impaired memory

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 420 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Change Detection in Over the Counter Medicine Labels | 60 minutes
  Looks at differences between two sets of images of medicine labels and locates the change between two sets of labels.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Becker, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Becker MW, Kashy DA, Harben A, Venkatesan K, Rodriguez A, Kebede M, Martin B, Breslow R, Bix L. A novel strategy to optimize critical information on over the counter labels for older adults. Health Sci Rep. 2023 Jan 25;6(1):e1062. doi: 10.1002/hsr2.1062. eCollection 2023 Jan. PMID 36712813
- [Result] Martin BA, Breslow RM, Sims A, Harben AL, Bix L, Becker MW. Identifying over-the-counter information to prioritize for the purpose of reducing adverse drug reactions in older adults: A national survey of pharmacists. J Am Pharm Assoc (2003). 2022 Jan-Feb;62(1):167-175.e1. doi: 10.1016/j.japh.2021.08.019. Epub 2021 Aug 23. PMID 34503908
- [Result] Harben AL, Kashy DA, Esfahanian S, Liu L, Bix L, Becker MW. Using change detection to objectively evaluate whether novel over-the-counter drug labels can increase attention to critical health information among older adults. Cogn Res Princ Implic. 2021 May 26;6(1):40. doi: 10.1186/s41235-021-00307-z. PMID 34041617